CLINICAL TRIAL: NCT04351126
Title: Pathophysiology and Nature of Ovarian Hyperstimulation Syndrome (OHSS) as a Clinical Entity Could be Fully Explained and Effectively Managed as a State of Defective Mineralocorticoid Response
Brief Title: Management of Ovarian Hyperstimulation Syndrome as a State of Defective Mineralocorticoid Response
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ganin Fertility Center (Other)
Responsible Party: Principal Investigator, Muhammad saber mahmoud sayed zeafan, Principal Investigator, Ganin Fertility Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MSM-01
Record Dates: First submitted 2020-04-14; First posted 2020-04-17 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Ovarian Hyperstimulation Syndrome
Keywords: OHSS; Mineralocorticoid; aldosterone
MeSH Terms: conditions — Ovarian Hyperstimulation Syndrome | interventions — Bromocriptine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Other): patients at high risk for OHSS who are receiving conventional treatment either as a prophylaxis (in the form of bromocriptine) or as a management in case of developing OHSS (as continual bromocriptine and fluid monitoring and or paracentesis and or tube thoracostomy)
  Interventions: Drug: Bromocriptine
- treatment group (Experimental): patient who has developed OHSS while on conventional lines of management (as continual bromocriptine and fluid monitoring and or paracentesis and or tube thoracostomy) patients in this group, fludrocortisone was added to conventional lines of management.
  Interventions: Drug: Fludrocortisone 0.1 Milligrams (mg); Drug: Bromocriptine
- prevention group (Experimental): patients at high risk for OHSS who are receiving fludrocortisone as a prophylaxis
  Interventions: Drug: Fludrocortisone 0.1 Milligrams (mg)

INTERVENTIONS:
Drug: Fludrocortisone 0.1 Milligrams (mg) — 0.2-0.6 mg/day of fludrocortisone is prescribed
  Arms: prevention group; treatment group
Drug: Bromocriptine — 2.5 mg prescribed Vaginally twice daily
  Arms: Control group; treatment group

SUMMARY:
lines of evidence that support nature of ovarian hyperstimulation syndrome (OHSS) as "defective mineralocorticoid response" are cited, our hypothesis is tested clinically in both prophylaxis against and treatment of OHSS.

DETAILED DESCRIPTION:
several studies state significant correlation between OHSS and activation of Renin-angiotensin-aldosterone system (RAAS), degree of activation of RAAS correlates with severity of OHSS. In OHSS there is a cascade of events that mainly involves capillary leak with resultant fluid shift and electrolytes imbalance, these consequences are more pronounced - according to our hypothesis - due to inadequate mineralocorticoid response/activity in susceptible individuals in the settings of high progesterone levels with its antimineralocorticoid property, OHSS can be interpreted as a (mineralocorticoid deficiency crisis) and may effectively be treated as being so, so we conducted this study to test the hypothesis in both treatment and prevention of OHSS.

ELIGIBILITY:
Inclusion Criteria: patients undergoing ICSI who were considered at risk of developing OHSS:

* polycystic ovaries and/or previous history of OHSS, AMH > 40 pmol/L but patients were finally included in the study if serum E2 levels reached >3000 pg/ml on day of hCG trigger or at any stage of folliculometry
* age: 18-40

Exclusion Criteria:

* retrieval of less than 20 oocytes
* age less than 18 or above 40

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 107 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-02-25 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
duration of recovery | 10 days
  Time needed for full clinical recovery
prevention of OHSS occurrence | 21 days
  percentage of cases that has developed OHSS in both control and prevention groups

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad S Zeafan, MBBCH, Principal Investigator — Ganin Fertility Center; khaled M Elqusi, BSc, Principal Investigator — Ganin Fertility Center; Hossam Elattar, MBBCH, Principal Investigator — Ganin Fertility Center; Hosam Zaki, MSc, FRCOG, Study Director — Ganin Fertility Center
Locations (1):
- Ganin Fertility Center, Cairo, Maadi, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Navot D, Margalioth EJ, Laufer N, Birkenfeld A, Relou A, Rosler A, Schenker JG. Direct correlation between plasma renin activity and severity of the ovarian hyperstimulation syndrome. Fertil Steril. 1987 Jul;48(1):57-61. doi: 10.1016/s0015-0282(16)59290-5. PMID 2439386
- [Background] Delbaere A, Bergmann PJ, Englert Y. Features of the Renin-angiotensin system in ascites and pleural effusion during severe ovarian hyperstimulation syndrome. J Assist Reprod Genet. 1997 May;14(5):241-4. doi: 10.1007/BF02765823. PMID 9147235
- [Background] Gomez-Sanchez E, Gomez-Sanchez CE. The multifaceted mineralocorticoid receptor. Compr Physiol. 2014 Jul;4(3):965-94. doi: 10.1002/cphy.c130044. PMID 24944027
- [Background] Dunne FP, Barry DG, Ferriss JB, Grealy G, Murphy D. Changes in blood pressure during the normal menstrual cycle. Clin Sci (Lond). 1991 Oct;81(4):515-8. doi: 10.1042/cs0810515. PMID 1657498
- [Background] Ujioka T, Matsuura K, Kawano T, Okamura H. Role of progesterone in capillary permeability in hyperstimulated rats. Hum Reprod. 1997 Aug;12(8):1629-34. doi: 10.1093/humrep/12.8.1629. PMID 9308783
- [Background] Lainas T, Petsas G, Stavropoulou G, Alexopoulou E, Iliadis G, Minaretzis D. Administration of methylprednisolone to prevent severe ovarian hyperstimulation syndrome in patients undergoing in vitro fertilization. Fertil Steril. 2002 Sep;78(3):529-33. doi: 10.1016/s0015-0282(02)03290-9. PMID 12215328
- [Background] Kim MK, Won HJ, Shim SH, Cha DH, Yoon TK. Spontaneous ovarian hyperstimulation syndrome following a thawed embryo transfer cycle. Clin Exp Reprod Med. 2014 Sep;41(3):140-5. doi: 10.5653/cerm.2014.41.3.140. Epub 2014 Sep 30. PMID 25309860